CLINICAL TRIAL: NCT05682326
Title: An Integrated Pharmacokinetic and Safety Open-label Basket Trial of Daprodustat for the Treatment of Anemia Associated With Chronic Kidney Disease in Male and Female Children and Adolescents Aged 3 Months to Under 18 Years Requiring or Not Requiring Dialysis
Brief Title: Anemia Studies in CKD: Erythropoiesis Via a Novel PHI Daprodustat - Pediatric (ASCEND-P)
Acronym: ASCEND-P
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 214066
Record Dates: First submitted 2023-01-04; First posted 2023-01-12 (Actual); Results first posted 2025-11-10 (Actual); Last update posted 2025-11-10 (Actual); Status verified 2025-10

CONDITIONS: Anaemia
Keywords: Daprodustat; ASCEND-P; Anemia; Chronic kidney disease; Erythropoiesis stimulating agent; Dialysis; Non-dialysis; 214066; 212914
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic | interventions — GSK1278863

STUDY DESIGN:
Intervention Model Description: This is an open-label single arm trial, where all participants are on active treatment with daprodustat.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Daprodustat (Experimental): All participants will receive daprodustat for up to 52 weeks.
  Interventions: Drug: Daprodustat

INTERVENTIONS:
Drug: Daprodustat — Daprodustat will be administered up to Week 52.

SUMMARY:
This is an international, multicenter trial, evaluating pharmacokinetics (PK) (4 weeks), safety (52 weeks), and hemoglobin (Hgb) response (52 weeks) to daprodustat in children and adolescent participants with anemia associated with chronic kidney disease (CKD) incorporating 2 independent sub-trials (Non dialysis [ND] and Dialysis [D]). This study will enroll participants with anemia associated with CKD, in 2 distinct sub-populations differing only by their CKD stage and dialysis requirement (ND: CKD stage 3 to 5 not yet receiving dialysis and D: CKD stage 5d undergoing peritoneal dialysis [PD] or hemodialysis [HD]).

The maximum duration of the study will be approximately 60 weeks, including Screening period (up to 4 weeks), treatment period (52 weeks), and follow-up period (4 weeks).

Outcome measures are identical for the ND and D sub-trials, but will be separately assessed in each sub- trials, overall and within each age subgroups (12 to less than [<] 18 years, 6 to <12 years, 2 to <6 years, and 3 months to <2 years). Except for PK and dose change, which is within each age group only.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 3 months to less than (<)18 years of age.
* Anemia associated with CKD stage 3, 4, 5 (not on dialysis) or who have dialysis-dependent CKD, defined as Hgb 7.0 to 11.0 g/dL (if not using erythropoiesis stimulating agents [ESAs]) or Hgb 9.5 to 12.0 g/dL if using ESAs.
* Written informed consent or assent as appropriate.

Exclusion Criteria:

* Kidney transplant recipient with a functioning allograft.
* Scheduled for elective kidney transplantation within 3 months.
* Transferrin saturation (TSAT) < 20 percent (%), or Ferritin <25 nanogram (ng)/milliliter (mL).
* History of bone marrow aplasia or pure red cell aplasia.
* Active hemolysis.
* Other causes of anemia.
* Active gastrointestinal bleeding within the last 4 weeks.
* Active or previous malignancy within the last 2 years.
* Acute or chronic infection requiring antimicrobial therapy.
* History of significant thrombotic or thromboembolic events within the last 8 weeks.
* Heart failure (HF) New York Heart Association (NYHA) Class IV
* Uncontrolled hypertension.
* Alanine aminotransferase (ALT) >2× upper limit of normal (ULN), bilirubin >1.5× ULN (unless bilirubin is fractionated and direct bilirubin <35%), and cirrhosis or current unstable liver or biliary disease.

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2023-09-06 (Actual); Primary Completion 2024-10-18 (Actual); Study Completion 2025-03-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- Japan (3):
  - GSK Investigational Site, Aichi
  - GSK Investigational Site, Saitama
  - GSK Investigational Site, Tokyo
- GSK Investigational Site, Yangsan, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled into two sub-trials based on dialysis status under a master protocol. The non-dialysis (ND) sub-trial enrolled pediatric participants with anemia associated with chronic kidney disease (CKD) not yet requiring dialysis in non-US countries. The dialysis (D) sub-trial enrolled pediatric participants with anemia associated with CKD requiring dialysis in non-US countries. Recruitment was conducted separately for each sub-trial.
Pre-assignment Details: A total of 4 participants were enrolled. As pre-specified in protocol design, data for the 2 sub-trials (ND and D) have been presented in two arms for this study.
Groups:
- Participants Requiring Dialysis (D): Participants received daprodustat orally once daily (QD) from Day 1 up to 52 weeks in the dialysis sub-trial. The dose of daprodustat was adjusted, if required, one step at a time in the range of 1 to 24 milligram (mg), to maintain the target range for hemoglobin (Hgb) between 10 to 12 grams per deciliter (g/dL).
- Participants Not Yet Requiring Dialysis (ND): Participants received daprodustat orally once daily (QD) from Day 1 up to 52 weeks in the non-dialysis sub-trial. The dose of daprodustat was adjusted, if required, one step at a time in the range of 1 to 24 mg, to maintain the target range for hemoglobin (Hgb) between 10 to 12 grams per deciliter (g/dL).
Period: Overall Study
Arm/Group | Participants Requiring Dialysis (D) | Participants Not Yet Requiring Dialysis (ND)
Started | 2 | 2
Completed | 1 | 2
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Participants Requiring Dialysis (D): Participants received daprodustat orally once daily (QD) from Day 1 up to 52 weeks in the dialysis sub-trial. The dose of daprodustat was adjusted, if required, one step at a time in the range of 1 to 24 mg, to maintain the target range for hemoglobin (Hgb) between 10 to 12 grams per deciliter (g/dL).
- Total: Total of all reporting groups
Arm/Group | Participants Requiring Dialysis (D) | Participants Not Yet Requiring Dialysis (ND) | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Customized [Count of Participants; unit: Participants]
  12 to <18 years | 2 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 0 | 2 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — "All Other Races" category (Asian - East Asian Heritage and Asian - Japanese Heritage where 0<n<11) are combined into one category to maintain participant confidentiality and privacy.
  Participants
    All Other Races | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study intervention, whether or not considered related to the study intervention. SAEs are defined as any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires inpatient hospitalization or prolongation of existing hospitalization; results in persistent or significant disability/incapacity; is a congenital anomaly/birth defect; or other situations as per medical and scientific judgement of the Investigator.
Time Frame: Up to 56 weeks
Population: The analysis was performed on the Safety Set that included all participants who were enrolled and took at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Requiring Dialysis (D) | Participants Not Yet Requiring Dialysis (ND)
Number analyzed (Participants) | 2 | 2
Participants
  Any AEs | 2 | 2
  Any SAEs | 1 | 0

2. Primary Outcome: Number of Participants With Adverse Event of Special Interests (AESIs)
Description: AESIs are AEs of scientific interest specific to the drug class as per investigator assessment. AESI included: Death, Myocardial Infarction (MI), stroke, Heart Failure (HF), thromboembolic events, thrombosis of vascular access, Thrombosis and/or tissue ischemia secondary to excessive erythropoiesis, New diagnosis of hypertension or worsening of existing hypertension, Cancer related mortality and tumor progression and recurrence, Esophageal and gastric erosions. Number of participants with any AESIs have been presented.
Time Frame: Up to 56 weeks
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Requiring Dialysis (D) | Participants Not Yet Requiring Dialysis (ND)
Number analyzed (Participants) | 2 | 2
Participants | 0 | 0

3. Primary Outcome: Number of Participants With AEs Leading to Study Intervention Discontinuation
Description: All AEs leading to study intervention discontinuation were collected. Number of participants with any AEs leading to study intervention discontinuation have been presented
Time Frame: Up to 52 weeks
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Requiring Dialysis (D) | Participants Not Yet Requiring Dialysis (ND)
Number analyzed (Participants) | 2 | 2
Participants | 0 | 0

4. Secondary Outcome: Change From Baseline in Hematology Parameter: Hematocrit
Description: Blood samples were collected to analyze the hematology parameter: hematocrit. Baseline value was defined as the last non-missing value prior to the start date and time of the study medication (Day 1). Change from Baseline was calculated as the value at indicated time point minus the value at Baseline.
Time Frame: Baseline (Day 1), at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: Safety Set. Only those participants who were measured and analyzed (i.e., contributed data reported in the table) were included in the Overall Number of Participants Analyzed field. 'Number Analyzed' signifies participants evaluable for the specified time points.
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells in blood
Arm/Group | Participants Requiring Dialysis (D) | Participants Not Yet Requiring Dialysis (ND)
Number analyzed (Participants) | 1 | 2
Percentage of red blood cells in blood
  Week 4 | 0.0160 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0030 (0.03818)
  Week 8 | 0.0530 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0025 (0.03889)
  Week 12 | -0.0280 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0135 (0.01485)
  Week 16 | -0.0200 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.0185 (0.03889)
  Week 20 | 0.0000 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.0005 (0.01909)
  Week 24 | 0.0050 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0060 (0.02687)
  Week 28 | 0.0340 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.0050 (0.03536)
  Week 32: number analyzed (Participants) | 1 | 1
  Week 32 | 0.0350 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0370 (NA) — NA indicates that standard deviation could not be calculated for single participant
  Week 36 | 0.0070 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0095 (0.02333)
  Week 40 | -0.0220 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0270 (0.04667)
  Week 44 | -0.0020 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.0060 (0.03677)
  Week 48: number analyzed (Participants) | 0 | 2
  Week 48 |  | 0.0035 (0.01909)
  Week 52 | -0.0320 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0020 (0.01980)

5. Secondary Outcome: Change From Baseline in Hematology Parameter: Reticulocytes/Erythrocytes
Description: Blood samples were collected to analyze the hematology parameter: Reticulocytes/Erythrocytes. Baseline value was defined as the last non-missing value prior to the start date and time of the study medication (Day 1). Change from Baseline was calculated as the value at indicated time point minus the value at Baseline.
Time Frame: Baseline (Day 1), at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Ratio of Reticulocytes to Erythrocytes
Arm/Group | Participants Requiring Dialysis (D) | Participants Not Yet Requiring Dialysis (ND)
Number analyzed (Participants) | 1 | 2
Ratio of Reticulocytes to Erythrocytes
  Week 4 | 0.0080 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.0039 (0.00686)
  Week 8 | -0.0020 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0031 (0.00134)
  Week 12 | 0.0060 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.0012 (0.00594)
  Week 16 | 0.0100 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.0024 (0.00481)
  Week 20 | 0.0110 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0001 (0.00693)
  Week 24 | 0.0060 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.0020 (0.00700)
  Week 28 | 0.0040 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0007 (0.00467)
  Week 32: number analyzed (Participants) | 1 | 1
  Week 32 | 0.0030 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.0037 (NA) — NA indicates that standard deviation could not be calculated for single participant
  Week 36 | 0.0020 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0010 (0.00573)
  Week 40 | 0.0070 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.0020 (0.00849)
  Week 44 | 0.0100 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0010 (0.00714)
  Week 48: number analyzed (Participants) | 0 | 2
  Week 48 |  | 0.0026 (0.00771)
  Week 52 | 0.0040 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0018 (0.00453)

6. Secondary Outcome: Change From Baseline in Hematology Parameter: Erythrocytes
Description: Blood samples were collected to analyze the hematology parameter: Erythrocytes. Baseline value was defined as the last non-missing value prior to the start date and time of the study medication (Day 1). Change from Baseline was calculated as the value at indicated time point minus the value at Baseline.
Time Frame: Baseline (Day 1), at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Trillion cells per Liter (10^12 cells/L)
Arm/Group | Participants Requiring Dialysis (D) | Participants Not Yet Requiring Dialysis (ND)
Number analyzed (Participants) | 1 | 2
Trillion cells per Liter (10^12 cells/L)
  Week 4 | 0.130 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.060 (0.4243)
  Week 8 | 0.480 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.045 (0.4313)
  Week 12 | -0.350 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.060 (0.2546)
  Week 16 | -0.350 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.280 (0.5374)
  Week 20 | 0.010 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.050 (0.2970)
  Week 24 | 0.030 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.025 (0.3889)
  Week 28 | 0.250 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.095 (0.4879)
  Week 32: number analyzed (Participants) | 1 | 1
  Week 32 | 0.350 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.350 (NA) — NA indicates that standard deviation could not be calculated for single participant
  Week 36 | 0.030 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.050 (0.3111)
  Week 40 | -0.330 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.310 (0.4808)
  Week 44 | -0.260 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.080 (0.5515)
  Week 48: number analyzed (Participants) | 0 | 2
  Week 48 |  | -0.025 (0.2758)
  Week 52 | -0.490 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.050 (0.2687)

7. Secondary Outcome: Change From Baseline in Hematology Parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Leukocytes and Platelet Count
Description: Blood samples were collected to analyze the hematology parameters: Basophils, Eosinophils, Lymphocytes, Monocytes, Neutrophils, Leukocytes and Platelet count. Baseline value was defined as the last non-missing value prior to the start date and time of the study medication (Day 1). Change from Baseline was calculated as the value at indicated time point minus the value at Baseline.
Time Frame: Baseline (Day 1), at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Giga cells per Liter (10^9 cells/L)
Arm/Group | Participants Requiring Dialysis (D) | Participants Not Yet Requiring Dialysis (ND)
Number analyzed (Participants) | 1 | 2
Giga cells per Liter (10^9 cells/L)
  Basophils: Week 4 | 0.0120 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0007 (0.01509)
  Basophils: Week 8 | -0.0177 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0087 (0.01232)
  Basophils: Week 12 | -0.0011 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0093 (0.01312)
  Basophils: Week 16 | -0.0062 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.0038 (0.02292)
  Basophils: Week 20 | 0.0085 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0162 (0.02295)
  Basophils: Week 24 | -0.0044 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0066 (0.02353)
  Basophils: Week 28 | 0.0182 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0003 (0.01458)
  Basophils: Week 32: number analyzed (Participants) | 1 | 1
  Basophils: Week 32 | -0.0209 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0314 (NA) — NA indicates that standard deviation could not be calculated for single participant
  Basophils: Week 36 | -0.0091 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0051 (0.02139)
  Basophils: Week 40 | -0.0020 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0063 (0.00522)
  Basophils: Week 44 | -0.0091 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0001 (0.00017)
  Basophils: Week 48: number analyzed (Participants) | 0 | 2
  Basophils: Week 48 |  | 0.0059 (0.00833)
  Basophils: Week 52 | 0.0012 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.0001 (0.00008)
  Eosinophils: Week 4 | 0.0146 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.4193 (0.63542)
  Eosinophils: Week 8 | -0.0962 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.2385 (0.30899)
  Eosinophils: Week 12 | -0.0072 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.2547 (0.11973)
  Eosinophils: Week 16 | 0.0239 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.1184 (0.15326)
  Eosinophils: Week 20 | -0.0037 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0989 (0.13988)
  Eosinophils: Week 24 | 0.0203 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0698 (0.18356)
  Eosinophils: Week 28 | -0.0578 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0238 (0.07607)
  Eosinophils: Week 32: number analyzed (Participants) | 1 | 1
  Eosinophils: Week 32 | -0.1571 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.2913 (NA) — NA indicates that standard deviation could not be calculated for single participant
  Eosinophils: Week 36 | -0.0775 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0395 (0.14069)
  Eosinophils: Week 40 | -0.1208 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0357 (0.07683)
  Eosinophils: Week 44 | -0.0522 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0395 (0.02754)
  Eosinophils: Week 48: number analyzed (Participants) | 0 | 2
  Eosinophils: Week 48 |  | 0.1645 (0.10537)
  Eosinophils: Week 52 | -0.0628 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0390 (0.00136)
  Lymphocytes: Week 4 | 0.2799 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.2606 (0.01499)
  Lymphocytes: Week 8 | 0.4370 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.4114 (0.49299)
  Lymphocytes: Week 12 | -0.2165 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.2552 (0.57253)
  Lymphocytes: Week 16 | -0.2907 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.2009 (0.40885)
  Lymphocytes: Week 20 | 0.1325 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.3649 (0.58710)
  Lymphocytes: Week 24 | -0.1535 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.3050 (0.58684)
  Lymphocytes: Week 28 | 0.0289 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.2517 (0.50673)
  Lymphocytes: Week 32: number analyzed (Participants) | 1 | 1
  Lymphocytes: Week 32 | -1.1501 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.6357 (NA) — NA indicates that standard deviation could not be calculated for single participant
  Lymphocytes: Week 36 | 0.0581 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.4619 (1.00143)
  Lymphocytes: Week 40 | -0.2134 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.4961 (0.05108)
  Lymphocytes: Week 44 | 0.5638 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.4021 (0.50620)
  Lymphocytes: Week 48: number analyzed (Participants) | 0 | 2
  Lymphocytes: Week 48 |  | -0.1701 (0.33923)
  Lymphocytes: Week 52 | 0.4700 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.5256 (0.60026)
  Monocytes: Week 4 | 0.0408 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.0318 (0.03079)
  Monocytes: Week 8 | 0.1094 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0230 (0.15981)
  Monocytes: Week 12 | -0.0258 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0536 (0.01924)
  Monocytes: Week 16 | -0.0289 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0148 (0.00684)
  Monocytes: Week 20 | 0.0132 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.0307 (0.11217)
  Monocytes: Week 24 | -0.0404 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.0310 (0.04098)
  Monocytes: Week 28 | 0.0169 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.0314 (0.06868)
  Monocytes: Week 32: number analyzed (Participants) | 1 | 1
  Monocytes: Week 32 | -0.2902 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0410 (NA) — NA indicates that standard deviation could not be calculated for single participant
  Monocytes: Week 36 | -0.0410 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.0596 (0.01360)
  Monocytes: Week 40 | -0.0708 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0884 (0.20985)
  Monocytes: Week 44 | 0.0601 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.0110 (0.02690)
  Monocytes: Week 48: number analyzed (Participants) | 0 | 2
  Monocytes: Week 48 |  | 0.0492 (0.04132)
  Monocytes: Week 52 | 0.0164 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.0112 (0.01583)
  Neutrophils: Week 4 | -0.1973 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.1626 (0.16602)
  Neutrophils: Week 8 | -3.5926 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.4712 (1.43005)
  Neutrophils: Week 12 | -0.1094 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.4876 (0.20136)
  Neutrophils: Week 16 | -1.7681 (NA) — NA indicates that standard deviation could not be calculated for single participant | 1.3315 (1.27070)
  Neutrophils: Week 20 | -0.8705 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.0296 (0.38241)
  Neutrophils: Week 24 | -1.2919 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.2346 (0.30353)
  Neutrophils: Week 28 | 1.6839 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.1160 (0.33096)
  Neutrophils: Week 32: number analyzed (Participants) | 1 | 1
  Neutrophils: Week 32 | -5.3517 (NA) — NA indicates that standard deviation could not be calculated for single participant | 1.1306 (NA) — NA indicates that standard deviation could not be calculated for single participant
  Neutrophils: Week 36 | 1.2095 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.4269 (0.70272)
  Neutrophils: Week 40 | -0.2730 (NA) — NA indicates that standard deviation could not be calculated for single participant | 1.0158 (0.85667)
  Neutrophils: Week 44 | 0.5974 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0185 (0.11095)
  Neutrophils: Week 48: number analyzed (Participants) | 0 | 2
  Neutrophils: Week 48 |  | 0.3055 (0.11948)
  Neutrophils: Week 52 | -0.0248 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.6728 (0.91533)
  Leukocytes: Week 4 | 0.150 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.045 (0.7849)
  Leukocytes: Week 8 | -3.160 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.315 (2.4254)
  Leukocytes: Week 12 | -0.360 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.510 (0.5798)
  Leukocytes: Week 16 | -2.070 (NA) — NA indicates that standard deviation could not be calculated for single participant | 1.240 (0.6505)
  Leukocytes: Week 20 | -0.720 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.315 (1.2516)
  Leukocytes: Week 24 | -1.470 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.060 (1.1879)
  Leukocytes: Week 28 | 1.690 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.385 (1.0112)
  Leukocytes: Week 32: number analyzed (Participants) | 1 | 1
  Leukocytes: Week 32 | -6.970 (NA) — NA indicates that standard deviation could not be calculated for single participant | 2.130 (NA) — NA indicates that standard deviation could not be calculated for single participant
  Leukocytes: Week 36 | 1.140 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.070 (1.8809)
  Leukocytes: Week 40 | -0.680 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.605 (0.9970)
  Leukocytes: Week 44 | 1.160 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.390 (0.7212)
  Leukocytes: Week 48: number analyzed (Participants) | 0 | 2
  Leukocytes: Week 48 |  | 0.310 (0.4384)
  Leukocytes: Week 52 | 0.400 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.170 (0.3253)
  Platelet count: Week 4 | 16.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -30.0 (26.87)
  Platelet count: Week 8 | -31.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -41.5 (34.65)
  Platelet count: Week 12 | -11.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -32.0 (39.60)
  Platelet count: Week 16 | -5.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -47.0 (14.14)
  Platelet count: Week 20 | 5.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -39.5 (27.58)
  Platelet count: Week 24 | -11.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -10.0 (7.07)
  Platelet count: Week 28 | 10.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -14.5 (6.36)
  Platelet count: Week 32: number analyzed (Participants) | 1 | 1
  Platelet count: Week 32 | 6.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | 1.0 (NA) — NA indicates that standard deviation could not be calculated for single participant
  Platelet count: Week 36 | -4.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -25.0 (0.00)
  Platelet count: Week 40 | 23.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -18.5 (27.58)
  Platelet count: Week 44 | 28.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -7.5 (37.48)
  Platelet count: Week 48: number analyzed (Participants) | 0 | 2
  Platelet count: Week 48 |  | -36.0 (35.36)
  Platelet count: Week 52 | 30.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | 11.0 (65.05)

8. Secondary Outcome: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Volume
Description: Blood samples were collected to analyze the hematology parameter: Erythrocytes Mean Corpuscular Volume. Baseline value was defined as the last non-missing value prior to the start date and time of the study medication (Day 1). Change from Baseline was calculated as the value at indicated time point minus the value at Baseline.
Time Frame: Baseline (Day 1), at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Femtoliter (fL)
Arm/Group | Participants Requiring Dialysis (D) | Participants Not Yet Requiring Dialysis (ND)
Number analyzed (Participants) | 1 | 2
Femtoliter (fL)
  Week 4 | 1.00 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.45 (0.919)
  Week 8 | 2.10 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.35 (0.919)
  Week 12 | 1.00 (NA) — NA indicates that standard deviation could not be calculated for single participant | 2.00 (1.414)
  Week 16 | 3.10 (NA) — NA indicates that standard deviation could not be calculated for single participant | 1.15 (1.344)
  Week 20 | -0.20 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.85 (1.202)
  Week 24 | 0.60 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.95 (1.202)
  Week 28 | 2.60 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.70 (1.131)
  Week 32: number analyzed (Participants) | 1 | 1
  Week 32 | 0.80 (NA) — NA indicates that standard deviation could not be calculated for single participant | 1.90 (NA) — NA indicates that standard deviation could not be calculated for single participant
  Week 36 | 1.00 (NA) — NA indicates that standard deviation could not be calculated for single participant | 1.25 (0.495)
  Week 40 | 2.10 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.35 (1.626)
  Week 44 | 5.60 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.20 (1.980)
  Week 48: number analyzed (Participants) | 0 | 2
  Week 48 |  | 1.35 (0.778)
  Week 52 | 3.40 (NA) — NA indicates that standard deviation could not be calculated for single participant | 1.45 (0.495)

9. Secondary Outcome: Change From Baseline in Hematology Parameter: Erythrocytes Mean Corpuscular Hemoglobin
Description: Blood samples were collected to analyze the hematology parameter: Erythrocytes Mean Corpuscular Hemoglobin. Baseline value was defined as the last non-missing value prior to the start date and time of the study medication (Day 1). Change from Baseline was calculated as the value at indicated time point minus the value at Baseline.
Time Frame: Baseline (Day 1), at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Picogram (pg)
Arm/Group | Participants Requiring Dialysis (D) | Participants Not Yet Requiring Dialysis (ND)
Number analyzed (Participants) | 1 | 2
Picogram (pg)
  Week 4 | 0.30 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.00 (0.849)
  Week 8 | 0.20 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.45 (0.071)
  Week 12 | 0.70 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.70 (0.141)
  Week 16 | 1.30 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.95 (0.212)
  Week 20 | 0.90 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.85 (0.212)
  Week 24 | 1.30 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.70 (0.000)
  Week 28 | 1.20 (NA) — NA indicates that standard deviation could not be calculated for single participant | 1.45 (0.212)
  Week 32: number analyzed (Participants) | 1 | 1
  Week 32 | 1.00 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.40 (NA) — NA indicates that standard deviation could not be calculated for single participant
  Week 36 | 0.50 (NA) — NA indicates that standard deviation could not be calculated for single participant | 1.15 (0.636)
  Week 40 | 1.60 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.55 (0.212)
  Week 44 | 2.10 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.55 (1.061)
  Week 48: number analyzed (Participants) | 0 | 2
  Week 48 |  | 0.80 (0.566)
  Week 52 | 1.80 (NA) — NA indicates that standard deviation could not be calculated for single participant | 1.95 (1.626)

10. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Calcium, Potassium, Sodium, Blood Urea Nitrogen (BUN)
Description: Blood samples were collected to analyze the clinical chemistry parameters: Calcium, Potassium, Sodium and BUN. Baseline value was defined as the last non-missing value prior to the start date and time of the study medication (Day 1). Change from Baseline was calculated as the value at indicated time point minus the value at Baseline.
Time Frame: Baseline (Day 1), at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: millimoles per liter (mmol/L)
Arm/Group | Participants Requiring Dialysis (D) | Participants Not Yet Requiring Dialysis (ND)
Number analyzed (Participants) | 1 | 2
millimoles per liter (mmol/L)
  Calcium: Week 4 | 0.0749 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.1123 (0.05293)
  Calcium: Week 8 | -0.1248 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.1248 (0.10585)
  Calcium: Week 12 | -0.0499 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.1372 (0.12350)
  Calcium: Week 16 | 0.0000 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.1372 (0.12350)
  Calcium: Week 20 | 0.0250 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.0873 (0.08821)
  Calcium: Week 24 | 0.0250 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.0873 (0.15878)
  Calcium: Week 28 | -0.0499 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.1871 (0.08821)
  Calcium: Week 32: number analyzed (Participants) | 1 | 1
  Calcium: Week 32 | 0.0250 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0000 (NA) — NA indicates that standard deviation could not be calculated for single participant
  Calcium: Week 36 | 0.1248 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.1372 (0.12350)
  Calcium: Week 40 | 0.0000 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.0624 (0.05293)
  Calcium: Week 44 | 0.1248 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.1248 (0.07057)
  Calcium: Week 48: number analyzed (Participants) | 0 | 2
  Calcium: Week 48 |  | -0.1123 (0.08821)
  Calcium: Week 52 | 0.0998 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.1747 (0.14114)
  Potassium: Week 4 | 0.40 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.35 (0.354)
  Potassium: Week 8 | 0.30 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.40 (0.000)
  Potassium: Week 12 | 0.40 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.30 (0.283)
  Potassium: Week 16 | 0.10 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.45 (0.212)
  Potassium: Week 20 | 0.30 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.10 (0.424)
  Potassium: Week 24 | 0.20 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.05 (0.495)
  Potassium: Week 28 | 0.30 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.55 (0.354)
  Potassium: Week 32: number analyzed (Participants) | 1 | 1
  Potassium: Week 32 | 0.30 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.30 (NA) — NA indicates that standard deviation could not be calculated for single participant
  Potassium: Week 36 | 0.20 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.35 (0.071)
  Potassium: Week 40 | 0.40 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.55 (0.354)
  Potassium: Week 44 | 0.20 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.40 (0.424)
  Potassium: Week 48: number analyzed (Participants) | 0 | 2
  Potassium: Week 48 |  | -0.25 (0.495)
  Potassium: Week 52 | 0.50 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.20 (0.283)
  Sodium: Week 4 | 0.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.5 (3.54)
  Sodium: Week 8 | 0.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.5 (0.71)
  Sodium: Week 12 | -1.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0 (0.00)
  Sodium: Week 16 | 0.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.5 (3.54)
  Sodium: Week 20 | 1.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -2.0 (2.83)
  Sodium: Week 24 | 0.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.5 (2.12)
  Sodium: Week 28 | -2.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.5 (3.54)
  Sodium: Week 32: number analyzed (Participants) | 1 | 1
  Sodium: Week 32 | 0.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -3.0 (NA) — NA indicates that standard deviation could not be calculated for single participant
  Sodium: Week 36 | 0.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.5 (2.12)
  Sodium: Week 40 | 0.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -2.5 (3.54)
  Sodium: Week 44 | 1.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.5 (4.95)
  Sodium: Week 48: number analyzed (Participants) | 0 | 2
  Sodium: Week 48 |  | -1.0 (2.83)
  Sodium: Week 52 | -1.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.5 (2.12)
  BUN: Week 4 | 0.9996 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0893 (3.40790)
  BUN: Week 8 | -0.2142 (NA) — NA indicates that standard deviation could not be calculated for single participant | 2.1242 (4.06424)
  BUN: Week 12 | 1.7136 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.6962 (2.54961)
  BUN: Week 16 | 1.3923 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.1964 (4.77106)
  BUN: Week 20 | 0.7854 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.8390 (0.83304)
  BUN: Week 24 | 0.6069 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0000 (3.02925)
  BUN: Week 28 | 3.6057 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0893 (2.90303)
  BUN: Week 32: number analyzed (Participants) | 1 | 1
  BUN: Week 32 | 2.2134 (NA) — NA indicates that standard deviation could not be calculated for single participant | 1.4280 (NA) — NA indicates that standard deviation could not be calculated for single participant
  BUN: Week 36 | 4.1055 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.4820 (1.33792)
  BUN: Week 40 | -0.6426 (NA) — NA indicates that standard deviation could not be calculated for single participant | 4.1948 (7.19446)
  BUN: Week 44 | 2.2848 (NA) — NA indicates that standard deviation could not be calculated for single participant | 1.1603 (2.90303)
  BUN: Week 48: number analyzed (Participants) | 0 | 2
  BUN: Week 48 |  | 0.4463 (2.90303)
  BUN: Week 52 | 1.9278 (NA) — NA indicates that standard deviation could not be calculated for single participant | 1.1424 (4.94777)

11. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter: Creatinine
Description: Blood samples were collected to analyze the clinical chemistry parameter: Creatinine. Baseline value was defined as the last non-missing value prior to the start date and time of the study medication (Day 1). Change from Baseline was calculated as the value at indicated time point minus the value at Baseline.
Time Frame: Baseline (Day 1), at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: micromoles per Liter (µmol/L)
Arm/Group | Participants Requiring Dialysis (D) | Participants Not Yet Requiring Dialysis (ND)
Number analyzed (Participants) | 1 | 2
micromoles per Liter (µmol/L)
  Week 4 | 21.2160 (NA) — NA indicates that standard deviation could not be calculated for single participant | -3.0940 (5.62574)
  Week 8 | 139.6720 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.4420 (9.37624)
  Week 12 | -1.7680 (NA) — NA indicates that standard deviation could not be calculated for single participant | 3.9780 (10.62640)
  Week 16 | 4.4200 (NA) — NA indicates that standard deviation could not be calculated for single participant | 14.5860 (19.37755)
  Week 20 | -22.1000 (NA) — NA indicates that standard deviation could not be calculated for single participant | 12.3760 (6.25082)
  Week 24 | -5.3040 (NA) — NA indicates that standard deviation could not be calculated for single participant | 24.3100 (26.87854)
  Week 28 | 78.6760 (NA) — NA indicates that standard deviation could not be calculated for single participant | 13.7020 (13.12673)
  Week 32: number analyzed (Participants) | 1 | 1
  Week 32 | 83.9800 (NA) — NA indicates that standard deviation could not be calculated for single participant | 48.6200 (NA) — NA indicates that standard deviation could not be calculated for single participant
  Week 36 | 95.4720 (NA) — NA indicates that standard deviation could not be calculated for single participant | 32.2660 (45.63101)
  Week 40 | 100.7760 (NA) — NA indicates that standard deviation could not be calculated for single participant | 65.4160 (75.00989)
  Week 44 | 115.8040 (NA) — NA indicates that standard deviation could not be calculated for single participant | 49.5040 (57.50758)
  Week 48: number analyzed (Participants) | 0 | 2
  Week 48 |  | 56.1340 (65.63365)
  Week 52 | 151.1640 (NA) — NA indicates that standard deviation could not be calculated for single participant | 73.8140 (94.38744)

12. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Alanine Aminotransferase (ALT), Alkaline Phosphatase (ALP) and Aspartate Aminotransferase (AST)
Description: Blood samples were collected to analyze the clinical chemistry parameters: ALT, ALP and AST. Baseline value was defined as the last non-missing value prior to the start date and time of the study medication (Day 1). Change from Baseline was calculated as the value at indicated time point minus the value at Baseline.
Time Frame: Baseline (Day 1), at Weeks 4, 8, 12, 24, 32, 36, 40, 48, and 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: International units per liter
Arm/Group | Participants Requiring Dialysis (D) | Participants Not Yet Requiring Dialysis (ND)
Number analyzed (Participants) | 1 | 2
International units per liter
  ALT: Week 4 | 2.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -2.0 (0.00)
  ALT: Week 8 | 2.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -2.5 (0.71)
  ALT: Week 12 | 2.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -3.5 (0.71)
  ALT: Week 24 | 0.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -3.5 (2.12)
  ALT: Week 32: number analyzed (Participants) | 1 | 1
  ALT: Week 32 | 1.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -5.0 (NA) — NA indicates that standard deviation could not be calculated for single participant
  ALT: Week 36 | -1.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -1.0 (0.00)
  ALT: Week 40 | -2.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -3.5 (2.12)
  ALT: Week 48: number analyzed (Participants) | 0 | 2
  ALT: Week 48 |  | -0.5 (4.95)
  ALT: Week 52 | 0.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -4.5 (0.71)
  ALP: Week 4: number analyzed (Participants) | 1 | 1
  ALP: Week 4 | 34.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -29.0 (NA) — NA indicates that standard deviation could not be calculated for single participant
  ALP: Week 8: number analyzed (Participants) | 1 | 1
  ALP: Week 8 | 13.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | 77.0 (NA) — NA indicates that standard deviation could not be calculated for single participant
  ALP: Week 12: number analyzed (Participants) | 1 | 1
  ALP: Week 12 | 31.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | 123.0 (NA) — NA indicates that standard deviation could not be calculated for single participant
  ALP: Week 24: number analyzed (Participants) | 1 | 1
  ALP: Week 24 | 36.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | 23.0 (NA) — NA indicates that standard deviation could not be calculated for single participant
  ALP: Week 32: number analyzed (Participants) | 1 | 1
  ALP: Week 32 | 29.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | 141.0 (NA) — NA indicates that standard deviation could not be calculated for single participant
  ALP: Week 36: number analyzed (Participants) | 1 | 1
  ALP: Week 36 | 14.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | 113.0 (NA) — NA indicates that standard deviation could not be calculated for single participant
  ALP: Week 40: number analyzed (Participants) | 1 | 1
  ALP: Week 40 | 2.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | 100.0 (NA) — NA indicates that standard deviation could not be calculated for single participant
  ALP: Week 48: number analyzed (Participants) | 0 | 1
  ALP: Week 48 |  | 35.0 (NA) — NA indicates that standard deviation could not be calculated for single participant
  ALP: Week 52: number analyzed (Participants) | 1 | 1
  ALP: Week 52 | 2.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | 46.0 (NA) — NA indicates that standard deviation could not be calculated for single participant
  AST: Week 4 | 3.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -1.0 (1.41)
  AST: Week 8 | 5.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -1.0 (1.41)
  AST: Week 12 | 0.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -4.0 (2.83)
  AST: Week 24 | -1.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -5.5 (3.54)
  AST: Week 32: number analyzed (Participants) | 1 | 1
  AST: Week 32 | 1.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -4.0 (NA) — NA indicates that standard deviation could not be calculated for single participant
  AST: Week 36 | -2.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -2.5 (3.54)
  AST: Week 40 | -3.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -4.0 (4.24)
  AST: Week 48: number analyzed (Participants) | 0 | 2
  AST: Week 48 |  | -4.5 (4.95)
  AST: Week 52 | -2.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -6.0 (4.24)

13. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameters: Bilirubin and Direct Bilirubin
Description: Blood samples were collected to analyze the clinical chemistry parameters: Bilirubin and Direct Bilirubin. Baseline value was defined as the last non-missing value prior to the start date and time of the study medication (Day 1). Change from Baseline was calculated as the value at indicated time point minus the value at Baseline.
Time Frame: Baseline (Day 1), at Weeks 4, 8, 12, 24, 32, 36, 40, 48, and 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: micromoles per Liter (µmol/L)
Arm/Group | Participants Requiring Dialysis (D) | Participants Not Yet Requiring Dialysis (ND)
Number analyzed (Participants) | 1 | 2
micromoles per Liter (µmol/L)
  Bilirubin: Week 4 | 0.0000 (NA) — NA indicates that standard deviation could not be calculated for single participant | 1.1115 (1.57190)
  Bilirubin: Week 8 | 0.0000 (NA) — NA indicates that standard deviation could not be calculated for single participant | 1.5390 (2.17647)
  Bilirubin: Week 12 | 0.0000 (NA) — NA indicates that standard deviation could not be calculated for single participant | 3.4200 (4.83661)
  Bilirubin: Week 24 | -1.7100 (NA) — NA indicates that standard deviation could not be calculated for single participant | 4.9590 (2.17647)
  Bilirubin: Week 32: number analyzed (Participants) | 1 | 1
  Bilirubin: Week 32 | 0.0000 (NA) — NA indicates that standard deviation could not be calculated for single participant | 3.4200 (NA) — NA indicates that standard deviation could not be calculated for single participant
  Bilirubin: Week 36 | 0.0000 (NA) — NA indicates that standard deviation could not be calculated for single participant | 1.9665 (0.36275)
  Bilirubin: Week 40 | 0.0000 (NA) — NA indicates that standard deviation could not be calculated for single participant | 3.5910 (0.24183)
  Bilirubin: Week 48: number analyzed (Participants) | 0 | 2
  Bilirubin: Week 48 |  | -0.3420 (0.48366)
  Bilirubin: Week 52 | -1.7100 (NA) — NA indicates that standard deviation could not be calculated for single participant | 1.6245 (2.29739)
  Direct Bilirubin: Week 4 | 0.0000 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0000 (0.00000)
  Direct Bilirubin: Week 8 | 0.0000 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.1710 (0.24183)
  Direct Bilirubin: Week 12 | 0.0000 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.4275 (0.60458)
  Direct Bilirubin: Week 24 | 0.0000 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.4275 (0.60458)
  Direct Bilirubin: Week 32: number analyzed (Participants) | 1 | 1
  Direct Bilirubin: Week 32 | 0.0000 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0000 (NA) — NA indicates that standard deviation could not be calculated for single participant
  Direct Bilirubin: Week 36 | 0.0000 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0855 (0.12092)
  Direct Bilirubin: Week 40 | 0.0000 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0000 (0.00000)
  Direct Bilirubin: Week 48: number analyzed (Participants) | 0 | 2
  Direct Bilirubin: Week 48 |  | 0.0855 (0.12092)
  Direct Bilirubin: Week 52 | 0.0000 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0855 (0.12092)

14. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter: Protein
Description: Blood samples were collected to analyze the clinical chemistry parameter: Protein. Baseline value was defined as the last non-missing value prior to the start date and time of the study medication (Day 1). Change from Baseline was calculated as the value at indicated time point minus the value at Baseline.
Time Frame: Baseline (Day 1), at Weeks 4, 8, 12, 24, 32, 36, 40, 48, and 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Grams per liter
Arm/Group | Participants Requiring Dialysis (D) | Participants Not Yet Requiring Dialysis (ND)
Number analyzed (Participants) | 1 | 2
Grams per liter
  Week 4 | 6.00 (NA) — NA indicates that standard deviation could not be calculated for single participant | -2.30 (1.838)
  Week 8 | 5.00 (NA) — NA indicates that standard deviation could not be calculated for single participant | -1.85 (1.202)
  Week 12 | -1.00 (NA) — NA indicates that standard deviation could not be calculated for single participant | -2.65 (0.495)
  Week 24 | 2.00 (NA) — NA indicates that standard deviation could not be calculated for single participant | -1.45 (2.051)
  Week 32: number analyzed (Participants) | 1 | 1
  Week 32 | 4.00 (NA) — NA indicates that standard deviation could not be calculated for single participant | 2.00 (NA) — NA indicates that standard deviation could not be calculated for single participant
  Week 36 | 6.00 (NA) — NA indicates that standard deviation could not be calculated for single participant | -1.65 (3.748)
  Week 40 | 3.00 (NA) — NA indicates that standard deviation could not be calculated for single participant | 2.25 (5.303)
  Week 48: number analyzed (Participants) | 0 | 2
  Week 48 |  | 0.10 (2.687)
  Week 52 | 3.00 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.65 (2.333)

15. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter: Ferritin
Description: Blood samples were collected to analyze the clinical chemistry parameter: Ferritin. Baseline value was defined as the last non-missing value prior to the start date and time of the study medication (Day 1). Change from Baseline was calculated as the value at indicated time point minus the value at Baseline.
Time Frame: Baseline (Day 1), at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: micrograms per liter (µg/L)
Arm/Group | Participants Requiring Dialysis (D) | Participants Not Yet Requiring Dialysis (ND)
Number analyzed (Participants) | 1 | 2
micrograms per liter (µg/L)
  Week 4 | -32.00 (NA) — NA indicates that standard deviation could not be calculated for single participant | -12.60 (20.365)
  Week 8 | 167.00 (NA) — NA indicates that standard deviation could not be calculated for single participant | -17.30 (12.304)
  Week 12 | 28.00 (NA) — NA indicates that standard deviation could not be calculated for single participant | -23.30 (19.375)
  Week 16 | -29.00 (NA) — NA indicates that standard deviation could not be calculated for single participant | -24.95 (9.970)
  Week 20 | -35.00 (NA) — NA indicates that standard deviation could not be calculated for single participant | -28.50 (13.435)
  Week 24 | -33.00 (NA) — NA indicates that standard deviation could not be calculated for single participant | -26.95 (22.698)
  Week 28 | -36.00 (NA) — NA indicates that standard deviation could not be calculated for single participant | -27.65 (25.951)
  Week 32: number analyzed (Participants) | 1 | 1
  Week 32 | -14.00 (NA) — NA indicates that standard deviation could not be calculated for single participant | -22.00 (NA) — NA indicates that standard deviation could not be calculated for single participant
  Week 36 | 42.00 (NA) — NA indicates that standard deviation could not be calculated for single participant | -31.00 (12.728)
  Week 40 | 42.00 (NA) — NA indicates that standard deviation could not be calculated for single participant | -9.60 (37.335)
  Week 44 | 75.00 (NA) — NA indicates that standard deviation could not be calculated for single participant | -3.00 (59.397)
  Week 48: number analyzed (Participants) | 0 | 2
  Week 48 |  | -16.30 (50.487)
  Week 52 | 39.00 (NA) — NA indicates that standard deviation could not be calculated for single participant | -5.05 (56.498)

16. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter: Transferrin Saturation
Description: Blood samples were collected to analyze the clinical chemistry parameter: Transferrin saturation. Transferrin saturation is measured as a percentage, it is the ratio of serum iron and total iron-binding capacity, multiplied by 100. Baseline value was defined as the last non-missing value prior to the start date and time of the study medication (Day 1). Change from Baseline was calculated as the value at indicated time point minus the value at Baseline.
Time Frame: Baseline (Day 1), at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage (%) of transferrin saturation
Arm/Group | Participants Requiring Dialysis (D) | Participants Not Yet Requiring Dialysis (ND)
Number analyzed (Participants) | 1 | 2
Percentage (%) of transferrin saturation
  Week 4 | -6.900 (NA) — NA indicates that standard deviation could not be calculated for single participant | -14.990 (43.8548)
  Week 8 | -2.300 (NA) — NA indicates that standard deviation could not be calculated for single participant | 6.385 (7.6155)
  Week 12 | 6.500 (NA) — NA indicates that standard deviation could not be calculated for single participant | -18.245 (68.9500)
  Week 16 | -0.900 (NA) — NA indicates that standard deviation could not be calculated for single participant | -2.775 (4.5608)
  Week 20 | -3.600 (NA) — NA indicates that standard deviation could not be calculated for single participant | -18.500 (55.8614)
  Week 24 | -7.770 (NA) — NA indicates that standard deviation could not be calculated for single participant | -12.995 (55.1614)
  Week 28 | -6.900 (NA) — NA indicates that standard deviation could not be calculated for single participant | -29.050 (56.4978)
  Week 32: number analyzed (Participants) | 1 | 1
  Week 32 | -8.100 (NA) — NA indicates that standard deviation could not be calculated for single participant | -69.000 (NA) — NA indicates that standard deviation could not be calculated for single participant
  Week 36 | 3.100 (NA) — NA indicates that standard deviation could not be calculated for single participant | -31.620 (62.7628)
  Week 40 | 3.100 (NA) — NA indicates that standard deviation could not be calculated for single participant | -32.230 (52.0006)
  Week 44 | -7.600 (NA) — NA indicates that standard deviation could not be calculated for single participant | -27.305 (27.8529)
  Week 48: number analyzed (Participants) | 0 | 2
  Week 48 |  | -25.715 (28.6873)
  Week 52 | -1.500 (NA) — NA indicates that standard deviation could not be calculated for single participant | -7.520 (51.5905)

17. Secondary Outcome: Change From Baseline in Clinical Chemistry Parameter: Estimated Glomerular Filtration Rate
Description: Blood samples were collected to analyze the clinical chemistry parameter: Estimated Glomerular Filtration Rate. Baseline value was defined as the last non-missing value prior to the start date and time of the study medication (Day 1). Change from Baseline was calculated as the value at indicated time point minus the value at Baseline.
Time Frame: Baseline (Day 1), at Weeks 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mL per minute per 1.73 square meter
Arm/Group | Participants Requiring Dialysis (D) | Participants Not Yet Requiring Dialysis (ND)
Number analyzed (Participants) | 1 | 2
mL per minute per 1.73 square meter
  Week 4 | -0.380 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.615 (0.7990)
  Week 8 | -2.020 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.310 (2.4042)
  Week 12 | 0.040 (NA) — NA indicates that standard deviation could not be calculated for single participant | -1.095 (3.0335)
  Week 16 | -0.060 (NA) — NA indicates that standard deviation could not be calculated for single participant | -1.530 (2.0365)
  Week 20 | 0.440 (NA) — NA indicates that standard deviation could not be calculated for single participant | -1.740 (0.3253)
  Week 24 | 0.130 (NA) — NA indicates that standard deviation could not be calculated for single participant | -2.655 (2.3405)
  Week 28 | -0.930 (NA) — NA indicates that standard deviation could not be calculated for single participant | -1.200 (1.2445)
  Week 32: number analyzed (Participants) | 1 | 1
  Week 32 | -1.320 (NA) — NA indicates that standard deviation could not be calculated for single participant | -4.650 (NA) — NA indicates that standard deviation could not be calculated for single participant
  Week 36 | -1.460 (NA) — NA indicates that standard deviation could not be calculated for single participant | -2.370 (5.1053)
  Week 40 | -1.580 (NA) — NA indicates that standard deviation could not be calculated for single participant | -6.565 (4.3346)
  Week 44 | -1.770 (NA) — NA indicates that standard deviation could not be calculated for single participant | -4.855 (4.0800)
  Week 48: number analyzed (Participants) | 0 | 2
  Week 48 |  | -5.410 (4.4548)
  Week 52 | -2.260 (NA) — NA indicates that standard deviation could not be calculated for single participant | -5.935 (6.6539)

18. Secondary Outcome: Change From Baseline in Hematology Parameter: Prothrombin International Normalized Ratio
Description: Blood samples were collected to analyze the hematology parameter: Prothrombin International Normalized Ratio. It is used to assess the clotting ability of blood. Baseline value was defined as the last non-missing value prior to the start date and time of the study medication (Day 1). Change from Baseline was calculated as the value at indicated time point minus the value at Baseline.
Time Frame: Baseline (Day 1), at Weeks 4, 8, 12, 24, 32, 36, 40, 48, and 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Participants Requiring Dialysis (D) | Participants Not Yet Requiring Dialysis (ND)
Number analyzed (Participants) | 1 | 1
Ratio
  Week 4 | -0.010 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.010 (NA) — NA indicates that standard deviation could not be calculated for single participant
  Week 8 | -0.040 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.050 (NA) — NA indicates that standard deviation could not be calculated for single participant
  Week 12 | 0.010 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.030 (NA) — NA indicates that standard deviation could not be calculated for single participant
  Week 24 | -0.040 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.010 (NA) — NA indicates that standard deviation could not be calculated for single participant
  Week 32: number analyzed (Participants) | 1 | 0
  Week 32 | -0.010 (NA) — NA indicates that standard deviation could not be calculated for single participant |
  Week 36 | 0.010 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.020 (NA) — NA indicates that standard deviation could not be calculated for single participant
  Week 40 | 0.030 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.010 (NA) — NA indicates that standard deviation could not be calculated for single participant
  Week 48: number analyzed (Participants) | 0 | 1
  Week 48 |  | -0.010 (NA) — NA indicates that standard deviation could not be calculated for single participant
  Week 52 | 0.030 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.040 (NA) — NA indicates that standard deviation could not be calculated for single participant

19. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: Systolic and diastolic blood pressure (BP) were assessed using an appropriate size cuff preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions (e.g., television, cell phones). Baseline value was defined as the last non-missing value prior to the start date and time of the study medication (Day 1). Change from Baseline was calculated as the value at indicated time point minus the value at Baseline.
Time Frame: Baseline (Day 1), at Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Participants Requiring Dialysis (D) | Participants Not Yet Requiring Dialysis (ND)
Number analyzed (Participants) | 2 | 2
millimeters of mercury (mmHg)
  SBP: Week 2 | 11.5 (9.19) | -8.0 (11.31)
  SBP: Week 4: number analyzed (Participants) | 1 | 2
  SBP: Week 4 | 9.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | 3.5 (7.78)
  SBP: Week 8: number analyzed (Participants) | 1 | 2
  SBP: Week 8 | 6.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.5 (16.26)
  SBP: Week 12: number analyzed (Participants) | 1 | 2
  SBP: Week 12 | 0.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -9.5 (7.78)
  SBP: Week 16: number analyzed (Participants) | 1 | 2
  SBP: Week 16 | 2.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -8.5 (2.12)
  SBP: Week 20: number analyzed (Participants) | 1 | 2
  SBP: Week 20 | 8.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -7.5 (9.19)
  SBP: Week 24: number analyzed (Participants) | 1 | 2
  SBP: Week 24 | 25.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -7.0 (2.83)
  SBP: Week 28: number analyzed (Participants) | 1 | 2
  SBP: Week 28 | 17.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0 (19.80)
  SBP: Week 32: number analyzed (Participants) | 1 | 1
  SBP: Week 32 | 20.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | 20.0 (NA) — NA indicates that standard deviation could not be calculated for single participant
  SBP: Week 36: number analyzed (Participants) | 1 | 2
  SBP: Week 36 | 16.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | 2.5 (14.85)
  SBP: Week 40: number analyzed (Participants) | 1 | 2
  SBP: Week 40 | 10.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -1.0 (28.28)
  SBP: Week 44: number analyzed (Participants) | 1 | 2
  SBP: Week 44 | 7.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -5.5 (0.71)
  SBP: Week 48: number analyzed (Participants) | 0 | 2
  SBP: Week 48 |  | 4.0 (29.70)
  SBP: Week 52: number analyzed (Participants) | 1 | 2
  SBP: Week 52 | 4.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0 (16.97)
  DBP: Week 2 | 3.5 (2.12) | -7.5 (3.54)
  DBP: Week 4: number analyzed (Participants) | 1 | 2
  DBP: Week 4 | 19.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | 2.5 (14.85)
  DBP: Week 8: number analyzed (Participants) | 1 | 2
  DBP: Week 8 | 8.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -3.0 (2.83)
  DBP: Week 12: number analyzed (Participants) | 1 | 2
  DBP: Week 12 | -4.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -1.0 (1.41)
  DBP: Week 16: number analyzed (Participants) | 1 | 2
  DBP: Week 16 | 5.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -8.0 (0.00)
  DBP: Week 20: number analyzed (Participants) | 1 | 2
  DBP: Week 20 | 4.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -10.0 (9.90)
  DBP: Week 24: number analyzed (Participants) | 1 | 2
  DBP: Week 24 | 16.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -4.5 (10.61)
  DBP: Week 28: number analyzed (Participants) | 1 | 2
  DBP: Week 28 | 6.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | 4.0 (8.49)
  DBP: Week 32: number analyzed (Participants) | 2 | 1
  DBP: Week 32 | 8.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | 7.0 (NA) — NA indicates that standard deviation could not be calculated for single participant
  DBP: Week 36: number analyzed (Participants) | 1 | 2
  DBP: Week 36 | 11.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | 5.0 (4.24)
  DBP: Week 40: number analyzed (Participants) | 1 | 2
  DBP: Week 40 | 2.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0 (5.66)
  DBP: Week 44: number analyzed (Participants) | 1 | 2
  DBP: Week 44 | 11.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | 4.5 (0.71)
  DBP: Week 48: number analyzed (Participants) | 0 | 2
  DBP: Week 48 |  | -2.0 (0.00)
  DBP: Week 52: number analyzed (Participants) | 1 | 2
  DBP: Week 52 | 1.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -6.0 (1.41)

20. Secondary Outcome: Change From Baseline in Heart Rate (HR)
Description: Heart rate (HR) were assessed using an appropriate size cuff preceded by at least 5 minutes of rest for the participant in a quiet setting without distractions (e.g., television, cell phones). Baseline value was defined as the last non-missing value prior to the start date and time of the study medication (Day 1). Change from Baseline was calculated as the value at indicated time point minus the value at Baseline.
Time Frame: Baseline (Day 1), at Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: beats per minute (bpm)
Arm/Group | Participants Requiring Dialysis (D) | Participants Not Yet Requiring Dialysis (ND)
Number analyzed (Participants) | 2 | 2
beats per minute (bpm)
  Week 2 | -12.5 (9.19) | -9.0 (4.24)
  Week 4: number analyzed (Participants) | 1 | 2
  Week 4 | 2.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -2.0 (18.38)
  Week 8: number analyzed (Participants) | 1 | 2
  Week 8 | 15.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -8.0 (28.28)
  Week 12: number analyzed (Participants) | 1 | 2
  Week 12 | 5.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -11.0 (43.84)
  Week 16: number analyzed (Participants) | 1 | 2
  Week 16 | -10.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -12.0 (14.14)
  Week 20: number analyzed (Participants) | 1 | 2
  Week 20 | 0.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | 4.0 (14.14)
  Week 24: number analyzed (Participants) | 1 | 2
  Week 24 | 8.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | 5.5 (6.36)
  Week 28: number analyzed (Participants) | 1 | 2
  Week 28 | 14.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | 3.0 (5.66)
  Week 32: number analyzed (Participants) | 1 | 1
  Week 32 | 11.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -12.0 (NA) — NA indicates that standard deviation could not be calculated for single participant
  Week 36: number analyzed (Participants) | 1 | 2
  Week 36 | 1.00 (NA) — NA indicates that standard deviation could not be calculated for single participant | 3.5 (7.78)
  Week 40: number analyzed (Participants) | 1 | 1
  Week 40 | -1.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | 30.0 (NA) — NA indicates that standard deviation could not be calculated for single participant
  Week 44: number analyzed (Participants) | 1 | 2
  Week 44 | 12.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -3.5 (12.02)
  Week 48: number analyzed (Participants) | 0 | 2
  Week 48 |  | -17.5 (14.85)
  Week 52: number analyzed (Participants) | 1 | 2
  Week 52 | -3.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | 3.0 (1.41)

21. Secondary Outcome: Change From Baseline in Weight
Description: Weight readings in kilogram (kg) were collected. Baseline value was defined as the last non-missing value prior to the start date and time of the study medication (Day 1). Change from Baseline was calculated as the value at indicated time point minus the value at Baseline.
Time Frame: Baseline (Day 1), at Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: kilograms (Kg)
Arm/Group | Participants Requiring Dialysis (D) | Participants Not Yet Requiring Dialysis (ND)
Number analyzed (Participants) | 2 | 2
kilograms (Kg)
  Week 2 | -1.00 (0.141) | -0.70 (0.566)
  Week 4: number analyzed (Participants) | 1 | 2
  Week 4 | -1.80 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.25 (1.485)
  Week 8: number analyzed (Participants) | 1 | 2
  Week 8 | -2.40 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.40 (0.141)
  Week 12: number analyzed (Participants) | 1 | 2
  Week 12 | 1.20 (NA) — NA indicates that standard deviation could not be calculated for single participant | 1.00 (0.566)
  Week 16: number analyzed (Participants) | 1 | 2
  Week 16 | -0.50 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.60 (0.283)
  Week 20: number analyzed (Participants) | 1 | 2
  Week 20 | 2.20 | 0.70 (0.849)
  Week 24: number analyzed (Participants) | 1 | 2
  Week 24 | 2.00 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.45 (0.212)
  Week 28: number analyzed (Participants) | 1 | 2
  Week 28 | 1.70 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.80 (0.990)
  Week 32: number analyzed (Participants) | 1 | 1
  Week 32 | 1.00 (NA) — NA indicates that standard deviation could not be calculated for single participant | 1.90 (NA) — NA indicates that standard deviation could not be calculated for single participant
  Week 36: number analyzed (Participants) | 1 | 2
  Week 36 | 0.20 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.95 (1.768)
  Week 40: number analyzed (Participants) | 1 | 2
  Week 40 | 0.80 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.95 (1.061)
  Week 44: number analyzed (Participants) | 1 | 2
  Week 44 | 1.50 (NA) — NA indicates that standard deviation could not be calculated for single participant | 1.85 (0.495)
  Week 48: number analyzed (Participants) | 0 | 2
  Week 48 |  | 2.90 (0.000)
  Week 52: number analyzed (Participants) | 1 | 2
  Week 52 | 1.30 (NA) — NA indicates that standard deviation could not be calculated for single participant | 2.70 (0.000)

22. Secondary Outcome: Change From Baseline in Height
Description: Height readings in centimeters (cm) were collected. Baseline value was defined as the last non-missing value prior to the start date and time of the study medication (Day 1). Change from Baseline was calculated as the value at indicated time point minus the value at Baseline.
Time Frame: Baseline (Day 1), at Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: centimeters (cm)
Arm/Group | Participants Requiring Dialysis (D) | Participants Not Yet Requiring Dialysis (ND)
Number analyzed (Participants) | 2 | 2
centimeters (cm)
  Week 2 | -1.50 (2.121) | 0.85 (1.202)
  Week 4: number analyzed (Participants) | 1 | 2
  Week 4 | 0.00 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.95 (0.495)
  Week 8: number analyzed (Participants) | 1 | 2
  Week 8 | 0.00 (NA) — NA indicates that standard deviation could not be calculated for single participant | 1.20 (0.707)
  Week 12: number analyzed (Participants) | 1 | 2
  Week 12 | 0.00 (NA) — NA indicates that standard deviation could not be calculated for single participant | 2.65 (0.071)
  Week 16: number analyzed (Participants) | 1 | 2
  Week 16 | 0.10 (NA) — NA indicates that standard deviation could not be calculated for single participant | 1.85 (1.485)
  Week 20: number analyzed (Participants) | 1 | 2
  Week 20 | 0.30 (NA) — NA indicates that standard deviation could not be calculated for single participant | 3.35 (0.495)
  Week 24: number analyzed (Participants) | 1 | 2
  Week 24 | 0.30 (NA) — NA indicates that standard deviation could not be calculated for single participant | 3.70 (0.707)
  Week 28: number analyzed (Participants) | 1 | 2
  Week 28 | 1.00 (NA) — NA indicates that standard deviation could not be calculated for single participant | 4.60 (0.141)
  Week 32: number analyzed (Participants) | 1 | 1
  Week 32 | 0.80 (NA) — NA indicates that standard deviation could not be calculated for single participant | 5.30 (NA) — NA indicates that standard deviation could not be calculated for single participant
  Week 36: number analyzed (Participants) | 1 | 2
  Week 36 | 0.50 (NA) — NA indicates that standard deviation could not be calculated for single participant | 5.00 (1.131)
  Week 40: number analyzed (Participants) | 1 | 2
  Week 40 | 0.20 (NA) — NA indicates that standard deviation could not be calculated for single participant | 4.50 (2.546)
  Week 44: number analyzed (Participants) | 1 | 2
  Week 44 | 0.20 (NA) — NA indicates that standard deviation could not be calculated for single participant | 5.65 (2.192)
  Week 48: number analyzed (Participants) | 0 | 2
  Week 48 |  | 5.65 (2.192)
  Week 52: number analyzed (Participants) | 1 | 2
  Week 52 | -0.70 (NA) — NA indicates that standard deviation could not be calculated for single participant | 6.25 (2.333)

23. Secondary Outcome: Absolute Values of Hemoglobin (Hgb)
Description: Blood samples were collected from all participants for measurement of Hgb values in grams per deciliter (g/dL). Baseline value was defined as the last non-missing value prior to the start date and time of the study medication (Day 1). Hgb results of participants with intercurrent events were excluded from the summary.
Time Frame: Baseline (Day 1), at Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: grams per deciliter
Arm/Group | Participants Requiring Dialysis (D) | Participants Not Yet Requiring Dialysis (ND)
Number analyzed (Participants) | 2 | 2
grams per deciliter
  Baseline (Day 1) | 11.00 (0.424) | 11.35 (0.919)
  Week 2 | 10.85 (1.061) | 11.90 (0.990)
  Week 4: number analyzed (Participants) | 1 | 2
  Week 4 | 11.80 (NA) — NA indicates that standard deviation could not be calculated for single participant | 11.50 (0.566)
  Week 8: number analyzed (Participants) | 0 | 2
  Week 8 |  | 11.65 (0.212)
  Week 12: number analyzed (Participants) | 0 | 2
  Week 12 |  | 11.80 (0.283)
  Week 16: number analyzed (Participants) | 0 | 2
  Week 16 |  | 10.95 (0.495)
  Week 20: number analyzed (Participants) | 0 | 2
  Week 20 |  | 11.55 (0.212)
  Week 24: number analyzed (Participants) | 0 | 2
  Week 24 |  | 11.70 (0.141)
  Week 28: number analyzed (Participants) | 0 | 2
  Week 28 |  | 11.65 (0.354)
  Week 32: number analyzed (Participants) | 0 | 1
  Week 32 |  | 11.80 (NA) — NA indicates that standard deviation could not be calculated for single participant
  Week 36: number analyzed (Participants) | 0 | 2
  Week 36 |  | 11.95 (0.354)
  Week 40: number analyzed (Participants) | 0 | 1
  Week 40 |  | 12.10 (NA) — NA indicates that standard deviation could not be calculated for single participant
  Week 44: number analyzed (Participants) | 0 | 1
  Week 44 |  | 11.20 (NA) — NA indicates that standard deviation could not be calculated for single participant
  Week 48: number analyzed (Participants) | 0 | 1
  Week 48 |  | 11.90 (NA) — NA indicates that standard deviation could not be calculated for single participant
  Week 52: number analyzed (Participants) | 0 | 1
  Week 52 |  | 12.60 (NA) — NA indicates that standard deviation could not be calculated for single participant

24. Secondary Outcome: Change From Baseline in Hemoglobin (Hgb)
Description: Blood samples were collected from all participants for measurement of Hgb values in g/dL. Baseline value was defined as the last non-missing value prior to the start date and time of the study medication (Day 1). Change from Baseline was calculated as the value at indicated time point minus the value at Baseline. Hgb results of participants with intercurrent events were excluded from the summary.
Time Frame: Baseline (Day 1), at Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: grams per Liter
Arm/Group | Participants Requiring Dialysis (D) | Participants Not Yet Requiring Dialysis (ND)
Number analyzed (Participants) | 2 | 2
grams per Liter
  Week 2 | -0.15 (0.636) | 0.55 (0.071)
  Week 4: number analyzed (Participants) | 1 | 2
  Week 4 | 0.5 (NA) — NA indicates that standard deviation could not be calculated for single participant. | 0.15 (1.485)
  Week 8: number analyzed (Participants) | 0 | 2
  Week 8 |  | 0.30 (1.131)
  Week 12: number analyzed (Participants) | 0 | 2
  Week 12 |  | 0.45 (0.636)
  Week 16: number analyzed (Participants) | 0 | 2
  Week 16 |  | -0.40 (1.414)
  Week 20: number analyzed (Participants) | 0 | 2
  Week 20 |  | 0.20 (0.707)
  Week 24: number analyzed (Participants) | 0 | 2
  Week 24 |  | 0.35 (1.061)
  Week 28: number analyzed (Participants) | 0 | 2
  Week 28 |  | 0.30 (1.273)
  Week 32: number analyzed (Participants) | 0 | 1
  Week 32 |  | 1.10 (NA) — NA indicates that standard deviation could not be calculated for single participant.
  Week 36: number analyzed (Participants) | 0 | 2
  Week 36 |  | 0.60 (0.566)
  Week 40: number analyzed (Participants) | 0 | 1
  Week 40 |  | 0.10 (NA) — NA indicates that standard deviation could not be calculated for single participant.
  Week 44: number analyzed (Participants) | 0 | 1
  Week 44 |  | -0.80 (NA) — NA indicates that standard deviation could not be calculated for single participant.
  Week 48: number analyzed (Participants) | 0 | 1
  Week 48 |  | -0.10 (NA) — NA indicates that standard deviation could not be calculated for single participant.
  Week 52: number analyzed (Participants) | 0 | 1
  Week 52 |  | 0.60 (NA) — NA indicates that standard deviation could not be calculated for single participant.

25. Secondary Outcome: Number of Participants With Hgb Values Above, Below and Within the Target Range (10 to 12 g/dL)
Description: Number of participants with Hgb values above, below, and within the target range (10 to 12 g/dL) were assessed. Baseline assessment was defined as the last non-missing value prior to the start date and time of the study drug (Day 1). Hgb results of participants with intercurrent events were excluded from the summary.
Time Frame: Baseline (Day 1), at Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, and 52
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Requiring Dialysis (D) | Participants Not Yet Requiring Dialysis (ND)
Number analyzed (Participants) | 2 | 2
Participants
  Baseline (Day 1): Above Target Range | 0 | 0
  Baseline (Day 1): Within Target Range | 2 | 2
  Baseline (Day 1): Below Target Range | 0 | 0
  Week 2: Above Target Range | 0 | 1
  Week 2: Within Target Range | 2 | 1
  Week 2: Below Target Range | 0 | 0
  Week 4: number analyzed (Participants) | 1 | 2
  Week 4: Above Target Range | 0 | 0
  Week 4: Within Target Range | 1 | 2
  Week 4: Below Target Range | 0 | 0
  Week 8: number analyzed (Participants) | 0 | 2
  Week 8: Above Target Range |  | 0
  Week 8: Within Target Range |  | 2
  Week 8: Below Target Range |  | 0
  Week 12: number analyzed (Participants) | 0 | 2
  Week 12: Above Target Range |  | 0
  Week 12: Within Target Range |  | 2
  Week 12: Below Target Range |  | 0
  Week 16: number analyzed (Participants) | 0 | 2
  Week 16: Above Target Range |  | 0
  Week 16: Within Target Range |  | 2
  Week 16: Below Target Range |  | 0
  Week 20: number analyzed (Participants) | 0 | 2
  Week 20: Above Target Range |  | 0
  Week 20: Within Target Range |  | 2
  Week 20: Below Target Range |  | 0
  Week 24: number analyzed (Participants) | 0 | 2
  Week 24: Above Target Range |  | 0
  Week 24: Within Target Range |  | 2
  Week 24: Below Target Range |  | 0
  Week 28: number analyzed (Participants) | 0 | 2
  Week 28: Above Target Range |  | 0
  Week 28: Within Target Range |  | 2
  Week 28: Below Target Range |  | 0
  Week 32: number analyzed (Participants) | 0 | 1
  Week 32: Above Target Range |  | 0
  Week 32: Within Target Range |  | 1
  Week 32: Below Target Range |  | 0
  Week 36: number analyzed (Participants) | 0 | 2
  Week 36: Above Target Range |  | 1
  Week 36: Within Target Range |  | 1
  Week 36: Below Target Range |  | 0
  Week 40: number analyzed (Participants) | 0 | 1
  Week 40: Above Target Range |  | 1
  Week 40: Within Target Range |  | 0
  Week 40: Below Target Range |  | 0
  Week 44: number analyzed (Participants) | 0 | 1
  Week 44: Above Target Range |  | 0
  Week 44: Within Target Range |  | 1
  Week 44: Below Target Range |  | 0
  Week 48: number analyzed (Participants) | 0 | 1
  Week 48: Above Target Range |  | 0
  Week 48: Within Target Range |  | 1
  Week 48: Below Target Range |  | 0
  Week 52: number analyzed (Participants) | 0 | 1
  Week 52: Above Target Range |  | 1
  Week 52: Within Target Range |  | 0
  Week 52: Below Target Range |  | 0

26. Secondary Outcome: Change in Daprodustat Dose From Starting Dose at Each Study Time Point
Description: Daprodustat dose was adjusted, if required, one step at a time in the range of 1 to 24 mg, to maintain the target range for Hgb between 10 to 12 g/dL. Dose change values of daprodustat from starting dose at each study time point were calculated as dose level at indicated time point minus starting dose at Day 1 (Baseline).
Time Frame: Day 1 (Baseline), at Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Participants Requiring Dialysis (D) | Participants Not Yet Requiring Dialysis (ND)
Number analyzed (Participants) | 2 | 2
milligrams
  Week 2 | 0 (0) | -1 (1.41)
  Week 4: number analyzed (Participants) | 1 | 2
  Week 4 | 0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.5 (0.71)
  Week 8: number analyzed (Participants) | 1 | 2
  Week 8 | -6 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.5 (0.71)
  Week 12: number analyzed (Participants) | 1 | 2
  Week 12 | -2 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.5 (0.71)
  Week 16: number analyzed (Participants) | 1 | 2
  Week 16 | 0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.5 (0.71)
  Week 20: number analyzed (Participants) | 1 | 2
  Week 20 | 0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.5 (0.71)
  Week 24: number analyzed (Participants) | 1 | 2
  Week 24 | 0 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.5 (0.71)
  Week 28: number analyzed (Participants) | 1 | 2
  Week 28 | -2 (NA) — NA indicates that standard deviation could not be calculated for single participant | -0.5 (0.71)
  Week 32: number analyzed (Participants) | 1 | 1
  Week 32 | -6 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0 (NA) — NA indicates that standard deviation could not be calculated for single participant
  Week 36: number analyzed (Participants) | 1 | 2
  Week 36 | -4 (NA) — NA indicates that standard deviation could not be calculated for single participant | -1 (1.41)
  Week 40: number analyzed (Participants) | 1 | 2
  Week 40 | -4 (NA) — NA indicates that standard deviation could not be calculated for single participant | -2 (0)
  Week 44: number analyzed (Participants) | 1 | 2
  Week 44 | -4 (NA) — NA indicates that standard deviation could not be calculated for single participant | -1 (0)
  Week 48: number analyzed (Participants) | 0 | 1
  Week 48 |  | -1 (NA) — NA indicates that standard deviation could not be calculated for single participant

27. Secondary Outcome: Number of Participants With 0 to 10, or Greater Than (>) 10 Dose Adjustments
Description: Number of participants who required daprodustat dose adjustments form the starting dose were assessed. Data were categorized for number of participants who required no dose change (0 times) to 10 times and >10 times dose adjustments during the study.
Time Frame: Up to Week 52
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Requiring Dialysis (D) | Participants Not Yet Requiring Dialysis (ND)
Number analyzed (Participants) | 2 | 2
Participants
  No dose change (0 time) | 1 | 0
  1 time | 0 | 0
  2 times | 0 | 1
  3 times | 0 | 0
  4 times | 0 | 0
  5 times | 0 | 0
  6 times | 1 | 1
  7 times | 0 | 0
  8 times | 0 | 0
  9 times | 0 | 0
  10 times | 0 | 0
  >10 times | 0 | 0

28. Secondary Outcome: Daprodustat Dose at Each Study Time Point
Description: Mean and standard deviation of daprodustat dose received by participants at each study time point has been presented.
Time Frame: Baseline (Day 1), at Weeks 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, and 48
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: milligrams
Arm/Group | Participants Requiring Dialysis (D) | Participants Not Yet Requiring Dialysis (ND)
Number analyzed (Participants) | 2 | 2
milligrams
  Baseline (Day 1) | 6.0 (0.00) | 2.0 (0.00)
  Week 2 | 6.0 (0.00) | 1.0 (1.41)
  Week 4: number analyzed (Participants) | 1 | 2
  Week 4 | 6.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | 1.5 (0.71)
  Week 8: number analyzed (Participants) | 1 | 2
  Week 8 | 0.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | 1.5 (0.71)
  Week 12: number analyzed (Participants) | 1 | 2
  Week 12 | 4.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | 1.5 (0.71)
  Week 16: number analyzed (Participants) | 1 | 2
  Week 16 | 6.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | 1.5 (0.71)
  Week 20: number analyzed (Participants) | 1 | 2
  Week 20 | 6.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | 1.5 (0.71)
  Week 24: number analyzed (Participants) | 1 | 2
  Week 24 | 6.00 (NA) — NA indicates that standard deviation could not be calculated for single participant | 1.5 (0.71)
  Week 28: number analyzed (Participants) | 1 | 2
  Week 28 | 4.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | 1.5 (0.71)
  Week 32: number analyzed (Participants) | 1 | 1
  Week 32 | 0.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | 2.0 (NA) — NA indicates that standard deviation could not be calculated for single participant
  Week 36: number analyzed (Participants) | 1 | 2
  Week 36 | 2.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | 1.0 (1.41)
  Week 40: number analyzed (Participants) | 1 | 2
  Week 40 | 2.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | 0.0 (0.00)
  Week 44: number analyzed (Participants) | 1 | 2
  Week 44 | 2.0 (NA) — NA indicates that standard deviation could not be calculated for single participant | 1.0 (0.00)
  Week 48: number analyzed (Participants) | 0 | 1
  Week 48 |  | 1.0 (NA) — NA indicates that standard deviation could not be calculated for single participant

29. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Daprodustat
Description: Blood samples were collected for the plasma concentrations of daprodustat from which pharmacokinetic (PK) parameters were determined. Mean and standard deviation of daprodustat Cmax at steady state obtained via modeling in each sub-trial (requiring Dialysis and not yet requiring Dialysis).
Time Frame: Day 1: 1, 2 and 6 hours Post-dose; Week 2: Pre-dose and 1, 2 and 6 hours Post-dose
Population: The analysis was performed on the All Pharmacokinetic Set that included all participants in the Safety analysis who had at least 1 non-missing PK assessment (non-quantifiable values will be considered as non-missing values).
Measure: Mean (Standard Deviation); unit: Nanograms per milliliters (ng/mL)
Arm/Group | Participants Requiring Dialysis (D) | Participants Not Yet Requiring Dialysis (ND)
Number analyzed (Participants) | 2 | 2
Nanograms per milliliters (ng/mL) | 115.047 (3.854) | 19.447 (10.770)

30. Secondary Outcome: Area Under the Curve (AUC) at Steady State of Daprodustat
Description: Blood samples were collected for the plasma concentrations of daprodustat from which PK parameters were determined. Mean and standard deviation of daprodustat AUC at steady state obtained via modeling in each sub-trial (requiring Dialysis and not yet requiring Dialysis).
Time Frame: Day 1: 1, 2 and 6 hours Post-dose; Week 2: Pre-dose and 1, 2 and 6 hours Post-dose
Population: All Pharmacokinetic Set
Measure: Mean (Standard Deviation); unit: Hours*nanogram per milliliter (h*ng/mL)
Arm/Group | Participants Requiring Dialysis (D) | Participants Not Yet Requiring Dialysis (ND)
Number analyzed (Participants) | 2 | 2
Hours*nanogram per milliliter (h*ng/mL) | 185.379 (8.661) | 56.634 (6.009)

31. Secondary Outcome: Plasma Concentrations of Daprodustat and Metabolites at Pre-dose (Ctrough)
Description: Blood samples were collected for the plasma concentrations of daprodustat and metabolites from which PK parameters were determined. Mean and standard deviation of raw daprodustat and metabolites (GSK2391220, GSK2487818, GSK2506102, GSK2506104, GSK2531398 and GSK2531401) at steady state at pre-dose obtained via modeling in each sub-trial (requiring Dialysis and not yet requiring Dialysis).
Time Frame: Pre-dose on Week 2
Population: All Pharmacokinetic Set
Measure: Mean (Standard Deviation); unit: Nanograms per milliliters (ng/mL)
Arm/Group | Participants Requiring Dialysis (D) | Participants Not Yet Requiring Dialysis (ND)
Number analyzed (Participants) | 2 | 2
Nanograms per milliliters (ng/mL)
  Daprodustat | 0.4995 (0.3698) | NA (NA) — Data could not be calculated as the concentration values were below the lower limit of quantification
  GSK2391220 | 6.540 (2.206) | NA (NA) — Data could not be calculated as the concentration values were below the lower limit of quantification
  GSK2487818 | 0.869 (0.137) | NA (NA) — Data could not be calculated as the concentration values were below the lower limit of quantification
  GSK2506102 | 3.040 (0.424) | NA (NA) — Data could not be calculated as the concentration values were below the lower limit of quantification
  GSK2506104: number analyzed (Participants) | 2 | 1
  GSK2506104 | 10.55 (3.18) | 0.143 (NA) — Standard deviation could not be calculated as a single participant was analyzed
  GSK2531398 | 2.490 (0.184) | NA (NA) — Data could not be calculated as the concentration values were below the lower limit of quantification
  GSK2531401: number analyzed (Participants) | 2 | 1
  GSK2531401 | 11.25 (1.48) | 0.127 (NA) — Standard deviation could not be calculated as a single participant was analyzed

ADVERSE EVENTS:
Time Frame: All-cause mortality, serious adverse events (SAEs) and non-serious adverse events (Non-SAEs) were collected up to 56 weeks.
Description: All-cause mortality, SAEs and non-SAEs were reported for Safety Set which included participants who were enrolled and received at least one dose of study medication.
Arm/Group | Participants Requiring Dialysis (D) | Participants Not Yet Requiring Dialysis (ND)
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Requiring Dialysis (D) (N=2) | Participants Not Yet Requiring Dialysis (ND) (N=2)
Congenital uterine anomaly (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Participants Requiring Dialysis (D) (N=2) | Participants Not Yet Requiring Dialysis (ND) (N=2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (2)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Serum ferritin increased (Investigations) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-11-18): https://cdn.clinicaltrials.gov/large-docs/26/NCT05682326/Prot_002.pdf
  • Statistical Analysis Plan (2025-07-14): https://cdn.clinicaltrials.gov/large-docs/26/NCT05682326/SAP_001.pdf